CLINICAL TRIAL: NCT02135302
Title: A Phase 1, Open-Label Study to Assess the Single-Dose Pharmacokinetics of Eravacycline in Subjects With Impaired Hepatic Function and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-434-013
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Impaired Hepatic Function
Keywords: hepatic
MeSH Terms: interventions — eravacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impaired hepatic function (Experimental): A single 1.5 mg/kg dose of eravacycline will be administered intravenously on Day 1 as a 60 minute infusion to each hepatically impaired subject.
  Interventions: Drug: eravacycline
- Healthy subjects (Experimental): A single 1.5 mg/kg dose of eravacycline will be administered intravenously on Day 1 as a 60 minute infusion to each healthy subject.
  Interventions: Drug: eravacycline

INTERVENTIONS:
Drug: eravacycline — Eravacycline (TP-434) is a parenteral and oral antibiotic of the tetracycline class that is highly active in vitro and in established animal infection models against both nosocomial and community-acquired methicillin-susceptible or -resistant Staphylococcus aureus strains, vancomycin-susceptible or -resistant Enterococcus faecium and Enterococcus faecalis, and penicillin-susceptible or -resistant strains of Streptococcus pneumoniae. In addition, eravacycline is highly active against clinically important species of Enterobacteriaceae (including those isolates that produce extended-spectrum β-lactamases and/or are carbapenem-resistant), Acinetobacter baumannii, and anaerobes.
  Other Names: TP-434

SUMMARY:
This is a multi-center, open-label clinical study to assess the single-dose PK of eravacycline in subjects with hepatic impairment and healthy subjects conducted at approximately 3 sites in the United States. This study includes an up to 21-day Screening Period, a 5-day Treatment Period, and an End of Study Visit occurring approximately 2 weeks (± 2 days) after initiation of study drug administration. Approximately 24 subjects will be enrolled: 18 subjects with impaired hepatic function (6 subjects who meet the criteria for each of the 3 Child-Pugh categories of mild [5 - 6 points], moderate [7 - 9 points], and severe [10 - 15 points]) and 6 healthy subjects without hepatic impairment. Healthy subjects will be matched to hepatically impaired subjects in gender, age, and body mass index (BMI). All subjects will be administered a single IV dose of eravacycline (1.5 mg/kg).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged ≥18 years at Screening;
2. Eligible female subjects of childbearing potential with a non-sterilized male sexual partner must agree to use 2 medically accepted, effective methods of birth control (eg, hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) beginning >30 days prior to study drug administration and continuing until 7 days after the end of the study. Female subjects who are postmenopausal must have been postmenopausal for >1 year if they wish not to use contraceptives. If postmenopausal status is questionable, the subject's follicle-stimulating hormone level must be checked and must be elevated and consistent with postmenopausal levels (ie, >40 IU/L); otherwise these subjects must agree to use contraceptives listed above;
3. Male subjects with sexual partners of childbearing potential must agree to use a barrier contraceptive from the time of study drug administration through 7 days after the end of the study;
4. Female subjects of childbearing potential (including females with questionable postmenopausal status) must have a negative pregnancy test prior to dosing (Screening and Day -1);
5. Has a body mass index of 17 kg/m2 to 40 kg/m2, inclusive;
6. Has negative alcohol and illicit drug screens;
7. Has a negative screen for Human immunodeficiency virus (HIV);
8. Is able to understand and comply with study procedures and give written informed consent according to institutional and regulatory guidelines;

   Subjects with hepatic impairment:
9. Has a positive diagnosis of liver cirrhosis that has been stable for 2 months and is confirmed by imaging techniques, biopsy, or physical signs consistent with a clinical diagnosis of liver cirrhosis (eg, liver firmness to palpation, splenic enlargement, spider angiomata, palmar erythema, parotid hypertrophy, testicular atrophy, gynecomastia);
10. Subjects with hepatic impairment must be categorized in 1 of the following:

    * Mild hepatic impairment: has impaired but stable hepatic function as evidenced by Child-Pugh Clinical Assessment Score of 5-6 at both Screening and Day -1;
    * Moderate hepatic impairment: has impaired but stable hepatic function as evidenced by Child-Pugh Clinical Assessment Score of 7-9 at both Screening and Day -1; or
    * Severe hepatic impairment: has impaired but stable hepatic function as evidenced by Child-Pugh Clinical Assessment Score of 10-15 at both Screening and Day -1;

    Healthy subjects without hepatic impairment:
11. Must be in good health as determined by screening medical history, physical examination, vital signs, blood chemistry, hematology, glucose, and coagulation performance at Screening;
12. Has a negative screen for hepatitis B (HBV) and hepatitis C (HCV); and
13. Should be matched to a subject with hepatic impairment in gender, age, and BMI.

Exclusion Criteria:

1. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the course of the study;
2. Has a history or current evidence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, neurological, or psychiatric disease that may pose a significant safety risk or diminish a subject's ability to undergo all study procedures and assessments;
3. Evidence of renal impairment with a creatinine clearance of <50 mL/min/1.73m2 as measured by the Cockcroft Gault formula;
4. Use of another investigational drug or device within 30 days prior to receiving eravacycline (TP-434), or within at least 5 half-lives of the previous investigational drug, whichever is longer;
5. Has a history of alcoholism or drug abuse within 2 years prior to dosing;
6. Has a typical weekly alcohol consumption of 14 alcoholic drinks. One drink is defined as 1 glass of beer (approximately 10 oz to 12 oz) or 1 can (12 oz) of beer, 1 glass of wine (approximately 4 oz to 5 oz), or 1 glass of distilled spirits (hard liquor) containing 1 oz of the liquor (1 oz of liquid is approximately 30 mL);
7. Use of alcohol within 48 hours prior to dosing;
8. Has had a major surgical procedure within 3 months prior to administration of study drug;
9. Has known allergies to tetracycline antibiotic or related compounds, or a history of multiple adverse drug allergies of any origin;
10. Has inadequate venous access;
11. Donated >500 mL of blood within 2 months prior to Screening;
12. Has a change in dose or frequency of any new or chronic dose-adjusted prescription or non-prescription medication, including vitamins or herbal medications, within 7 days or 5 half-lives (if known), whichever is longer, within 2 weeks prior to dosing;
13. Is a member of the clinical site personnel directly affiliated with this study;
14. Has poor mental function or any other reason to expect subject difficulty in complying with the requirements of the study in the judgment of the investigator;
15. Fails to comply with protocol requirements, or whose further participation in the study would be unsuitable to the subject, as determined by the investigator;
16. Clinically significant abnormal electrocardiograms (ECGs) (QTcB or QTcF >500 msec);

    Subjects with hepatic impairment:
17. Has active HCV or HBV and is receiving antiviral therapy (either prescribed or herbal);
18. Has fluctuating or rapidly deteriorating hepatic function as indicated by clinical and/or laboratory signs of hepatic impairment (advanced ascites, infection of ascites, fever, or active gastrointestinal bleeding);
19. Has sodium levels 125 mmol/L;
20. Has platelets <40,000 × 109/L of blood or evidence of severe active or recent bleeding;
21. Has refractory encephalopathy, as judged by the investigator, or significant central nervous system disease (eg, dementia or seizures) which the investigator considers to interfere with informed consent, conduct, completion, or results of this study, or constitutes an unacceptable risk to the subject;
22. Has signs of active infection;
23. Has experienced esophageal variceal bleeding within the past 6 months;
24. Has a Transjugular Intrahepatic Portosystemic Shunt placement;

    Subjects without hepatic impairment:
25. Has aspartate aminotransferase or alanine aminotransferase >1.5 × upper limit of normal (ULN); alkaline phosphatase or bilirubin 1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination;
26. Has systolic blood pressure outside of the range of 90-160 mmHg, or diastolic blood pressure outside the range of 45-100 mmHg, or heart rate outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects;
27. Has a history of Gilbert's disease; or
28. Takes any concomitant medication, either prescribed or over-the-counter. This includes use of any prescription or non-prescription medication, including vitamins or herbal medications, within 7 days or 5 half-lives (if known), whichever is longer, prior to dosing and within 24 hours after dosing, excluding hormonal contraceptives. The use of acetaminophen, naproxen, and ibuprofen is permitted except for within 24 hours prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
This study is being conducted to assess the pharmacokinetic (PK) profile of eravacycline | one year
  To assess the pharmacokinetic (PK) profile of eravacycline after administration of a single intravenous (IV) dose (1.5 mg/kg) to subjects with mild, moderate, and severe impaired hepatic function compared with normal healthy subjects

SECONDARY OUTCOMES:
Safety and tolerability of Eravacycline | one year
  To determine the safety and tolerability of eravacycline after administration of a single IV dose (1.5 mg/kg) in subjects with mild, moderate, and severe impaired hepatic function compared with normal healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Principal Investigator — New Orleans Center for Clinical Research; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Chris Galloway, MD, Principal Investigator — Davia Clinical Research
Locations (3):
- United States (3):
  - Davita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center for Clinical Research, Knoxville, Tennessee